CLINICAL TRIAL: NCT00129168
Title: An Open-Label, Phase I/II, Multicenter Dose Escalation Study of Zosuquidar, Daunorubicin, and Cytarabine in Patients Ages 55-75 With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Zosuquidar in Combination With Daunorubicin and Cytarabine in Patients Ages 55-75 With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kanisa Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAN-979-01
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Leukemia, Myeloid
Keywords: Leukemia, Myeloid; Relapse; Chemotherapy; Zosuquidar; Daunorubicin; Cytarabine; Acute; AML; Adult AML
MeSH Terms: conditions — Leukemia, Myeloid; Recurrence; Leukemia, Myeloid, Acute | interventions — zosuquidar trihydrochloride; Daunorubicin; Cytarabine

INTERVENTIONS:
Drug: Zosuquidar
Drug: Daunorubicin
Drug: Cytarabine

SUMMARY:
Chemotherapy drugs use different ways to stop cancer cells from dividing so they stop growing or die. Zosuquidar may help daunorubicin and cytarabine kill more cancer cells by making cancer cells more sensitive to the drugs. It is not yet known whether daunorubicin and cytarabine are more effective with or without zosuquidar in treating acute myeloid leukemia.

DETAILED DESCRIPTION:
Purpose:

Phase I:

To Evaluate the safety of different doses of zosuquidar.

Phase II:

This study is designed to study the safety and effectiveness of zosuquidar when given with daunorubicin and cytarabine in newly diagnosed AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute myeloid leukemia
* Ages 55-75 years

Exclusion Criteria:

* Acute promyelocytic leukemia (FAB M3)
* Patients must not have received prior chemotherapy for AML.
* Prior exposure to anthracycline
* Use of any investigational agent within 4 weeks prior to enrollment into the study

For Phase II:

* Patients must be P-glycoprotein positive

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

REFERENCES:
- [Derived] Marcelletti JF, Sikic BI. Continuous 72-h infusion of zosuquidar with chemotherapy in patients with newly diagnosed acute myeloid leukemia stratified for leukemic blast P-glycoprotein phenotype. Cancer Chemother Pharmacol. 2024 Jun;93(6):595-604. doi: 10.1007/s00280-024-04656-6. Epub 2024 Feb 26. PMID 38407601